CLINICAL TRIAL: NCT02142322
Title: A Phase II Trial of Perioperative Chemotherapy With Oxaliplatin, 5-Fluorouracil, Leucovorin(MODIFIED FOLFOX6) in Patients With Locally Advanced Operable Gastric Cancer
Brief Title: Perioperative mFOLFOX-6 in Locally Advanced Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seock-Ah Im, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-0406-127-007
Record Dates: First submitted 2011-06-28; First posted 2014-05-20 (Estimated); Last update posted 2025-04-17 (Actual); Status verified 2014-05

CONDITIONS: Advanced Gastric Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Modified FOLFOX6 (Experimental): Modified FOLFOX6 regimen consists of oxaliplatin 100 mg/m2 and FA 100 mg/m2 given as a 2 hour intravenous infusion, followed by 5-FU 2.4 g/m2 given as a continuous infusion over 46 hour, repeated every 2 weeks. Patients receive 4 cycles of neoadjuvant modified FOLFOX6 followed by curative radical surgery with D2 dissection and 4 cycles of adjuvant modified FOLFOX6.
  Interventions: Drug: MODIFIED FOLFOX6

INTERVENTIONS:
Drug: MODIFIED FOLFOX6 — Modified FOLFOX6 regimen consists of oxaliplatin 100 mg/m2 and FA 100 mg/m2 given as a 2 hour intravenous infusion, followed by 5-FU 2.4 g/m2 given as a continuous infusion over 46 hour, repeated every 2 weeks. Patients receive 4 cycles of neoadjuvant modified FOLFOX6 followed by curative radical surgery with D2 dissection and 4 cycles of adjuvant modified FOLFOX6.

SUMMARY:
This is a Phase II Trial of Perioperative Chemotherapy with Oxaliplatin, 5-Fluorouracil, Leucovorin(MODIFIED FOLFOX6)in Patients with Locally Advanced Operable Gastric Cancer.

DETAILED DESCRIPTION:
The main purpose of this study is to evaluate response rate (clinical response and pathological response) of oxaliplatin, 5-fluorouracil, leucovorin(MODIFIED FOLFOX6)

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated patients with pathologically proven advanced gastric adenocarcinoma with regional LN metastasis are eligible for this study (clinical stage: cT2-4 and N+). At least one measurable regional lymph node metastasis according to the Response Evaluation Criteria in Solid Tumors (RECIST v. 1.0) [17] is required. Other eligibility criteria include age between 18 and 75 years, Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1, no prior chemotherapy or radiotherapy, and adequate bone marrow, hepatic and renal function (absolute neutrophil count [ANC] ≥ 1.5ⅹ109/L, platelet count ≥ 100ⅹ109/L, total bilirubin ≤ 1.5ⅹupper limit of normal [ULN], serum transaminases ≤ 2.5ⅹULN, alkaline phosphatase ≤ 2.5ⅹULN, serum creatinine ≤ 1.5ⅹULN or actual or calculated creatinine clearance ≥ 50 mL/min).

Exclusion Criteria:

* Exclusion criteria include clinical stage T1 tumors, clinical or radiologic evidence of distant metastasis, intestinal obstruction or impending obstruction, active tumor bleeding, interstitial pneumonitis or symptomatic pulmonary fibrosis, peripheral neuropathy of National Cancer Institute Common Toxicity Criteria (NCI-CTC) grade ≥1, pregnant or breastfeeding patients, and other serious diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2004-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
response rate | 22 weeks
  response rate by the RECIST criteria

SECONDARY OUTCOMES:
Grade 3-4 toxicity | one year
  toxicity : Grade 3-4 toxicity by the NCI-CTCAE v3.0
median overall survival | 1 year
  median value of the time from enrollment to the patient's death
median time to treatment failure | 1 year
  median value of the time from enrollment to disease progression, withdrawl of consent, or unacceptable toxicity
resection rate | 1 year
  the rate of patients whose tumor was completely resected

CONTACTS AND LOCATIONS:
Overall Officials: Seock-Ah Im, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul